CLINICAL TRIAL: NCT06820112
Title: This Study Retrospectively Collected Relevant Patient Data to Compare the Effects of Different Respiratory Support Modalities in Patients With Acute Pulmonary Edema.
Brief Title: Comparison of Respiratory Support for Acute Pulmonary Edema
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Qiaoyun Huang, Dr., The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 20252502
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Edema - Acute
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oxygen therapy
  Interventions: Other: mechanical ventilation

INTERVENTIONS:
Other: mechanical ventilation — patients who received mechanical ventilation

SUMMARY:
This study is a retrospective study. The demographic and vital signs of patients with acute pulmonary edema are retrospectively collected to compare the prognosis of patients after receiving different respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute pulmonary edema

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with acute pulmonary edema
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-06 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
death rate | 28 days

IPD SHARING:
Plan to Share IPD: No